CLINICAL TRIAL: NCT07028671
Title: Exploratory Pilot Investigation of Motilium's Effectiveness and Safety for the OTC Treatment of Dyspepsia-related Symptoms Among Chinese Suffers Using Real-world Evidence: A Non-interventional, Prospective, Observational Study
Brief Title: Exploratory Investigation of Motilium's Effectiveness and Safety for the OTC Treatment of Dyspepsia-related Symptoms
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Other Study IDs: R033812GAI4001
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to understand the effectiveness and safety of Motilium among study participants with dyspepsia-related symptoms in real-world settings in China.

ELIGIBILITY:
Inclusion Criteria:

* Individuals purchased OTC Motilium at pharmacies for themselves for the treatment of one or more dyspepsia-related symptoms including postprandial fullness, early satiation, epigastric pain, epigastric burning, belching, epigastric bloating, nausea, and vomiting
* Provided signed and dated informed consent

Exclusion Criteria:

* Individuals who suffered from dyspepsia-related symptoms ≥ 3 days/week for at least 3 months prior to joining the study
* Individuals who suffered exclusively from heartburn
* Individuals taking or planning to take dyspepsia-related medication, including but not limited to proton pump inhibitors, hydrotalcite, Talcid, Sanjiu Weitai, JianWeiXiaoShiPian, Jiangzhong Jianwei, Digestive enzyme, Itopride, Mosapride, and Famotidine
* History of, or current, cardiac disease or cardiac arrhythmias including QT prolongation, ventricular tachycardia, ventricular fibrillation and Torsades de Pointes
* Any of the following warning signs: black stool, unintended weight loss, progressive dysphagia, persistent vomiting, abdominal mass, and fever
* Diagnosed with accompanying GI or other disease (e.g., GI tumors, peptic ulcer, and hiatal hernia)
* Conditions with elevated health risk if having increased gastric motility (e.g., GI hemorrhage, mechanical obstruction or perforation)
* Hepatic dysfunction and renal insufficiency
* Concomitant use with oral ketoconazole, erythromycin, or other potent inhibitors of CYP3A4 enzymes that may prolong the QTc interval (refer to Chinese OTC label. e.g., fluconazole, voriconazole, clarithromycin, amiodarone, telithromycin, itraconazole, posaconazole, ritonavir, saquinavir, and telaprevir)
* Known allergies to Motilium (domperidone) or any other ingredient of Motilium
* Pregnant, breast feeding female or planning to become pregnant (either potential participant or potential participant's partner)
* Individuals who are currently taking Motilium
* Individuals who did not get relieved from dyspepsia-related symptoms after taking Motilium
* Individuals participating in any other clinical trials during this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study participant recruitment will occur at retail pharmacies in different provinces across China. Consumers assessed in this study are adult participants who purchase OTC Motilium at pharmacies to treat dyspepsia-related symptoms in China. Consumers who fulfill the pre-defined inclusion and exclusion criterion and sign the informed consent form are study participants. The decision of individuals to participate in this study must not, in any way, impact upon the standard of care that they are receiving or any benefits to which they are otherwise entitled. The treatment decision must have been taken prior to and independently of the patient's inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Motilium | Day 7
  To evaluate the effectiveness of Motilium for treating dyspepsia-related symptoms among adult study participants who purchase OTC Motilium in China
Safety of Motilium | Day 7
  To evaluate safety of treatments, based on adverse event (AE) reporting throughout the study period

OTHER OUTCOMES:
Overall treatment effect (OTE) with "improved significantly" or "improved" | Day 3
  Proportion of participants who were classified as responders (overall treatment effect (OTE) with "improved significantly" or "improved") on Day 3 or earlier if the treatment is < 3 days regardless of whether or not they were continuing use Motilium
Overall treatment effect (OTE) with "improved significantly" or "improved" | Day 7
  Proportion of participants who were classified as responders (OTE with "improved significantly" or "improved") on Day 7 or earlier if the treatment is < 7 days regardless of whether or not they were continuing use Motilium
Change in individual symptom GOS score≥ 2 | Day 3 and 7
  Proportion of participants with a change in individual symptom GOS score (ΔGOS) ≥ 2 within first 3 days and first 7 days compared to baseline for each symptom (i.e., postprandial fullness, early satiation, epigastric pain, epigastric burning, belching, epigastric bloating, nausea, and vomiting)
Time to change in Global Overall Symptom (GOS) ≥ 2 | Day 7
  Time to ≥ 2-point change in GOS score (ΔGOS)
Participants with improvement in GOS score | Day 3 and 7
  Proportion of participants with a change in individual symptom GOS score (ΔGOS) ≥ 2 within first 3 days and first 7 days compared to baseline for each symptom (i.e., postprandial fullness, early satiation, epigastric pain, epigastric burning, belching, epigastric bloating, nausea, and vomiting)
Participants with improvement in GOS score ≥ 2 | Day 7
  Proportion of participants with improvement in GOS score (ΔGOS) ≥ 2 and sustained without worsening for the rest of study period compared with baseline
Participants with improvement in individual symptoms using GOS score ≥ 2 | Day 7
  Proportion of participants with improvement in individual symptoms using GOS score
  ≥ 2 and sustained without worsening for the rest of study period compared to baseline of that specific symptom (i.e., postprandial fullness, early satiation, epigastric pain, epigastric burning, belching, epigastric bloating, nausea, and vomiting)
Positive feedback of the treatment | Day 7
  Proportion of participants who have positive satisfaction of treatment (Somewhat satisfied or Very satisfied)
Severity of AE and Serious Adverse Event (SAE) | Day 7
  Incidence and severity of AE and Serious Adverse Event (SAE) during the observational period
Took Motilium three times a day | Day 7
  Proportion of participants who took Motilium three times a day during treatment period
Took Motilium frequency | Day 7
  Proportion of participants who took Motilium for 1, 2, 3, 4, 5, 6, and 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jie Liu, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No